CLINICAL TRIAL: NCT04293094
Title: A Phase 1, Multicenter, Open-label, Dose-Exploration and Dose-Expansion Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Efficacy of AMG 650 in Subjects With Advanced Solid Tumors
Brief Title: Study of AMG 650 in Adult Participants With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Volastra Therapeutics, Inc. (Industry)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20190131
Record Dates: First submitted 2020-03-02; First posted 2020-03-03 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Advanced Solid Tumors
Keywords: AMG 650; Locally-advanced/metastatic solid tumors; p53 mutation; Serous like endometrial cancers; Triple negative breast cancer (TNBC); High grade serous ovarian cancer (HGSOC)
MeSH Terms: conditions — Triple Negative Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose Exploration Phase (Experimental): Participants will receive AMG 650 in 1 of 3 alternative schedules. The maximum tolerated dose (MTD) of each schedule will be estimated using isotonic regression (Ji et al, 2010). The Recommended Phase 2 Dose (RP2D) may be identified based on emerging safety, efficacy, and pharmacodynamics (PD) data prior to reaching an MTD.
  Interventions: Drug: AMG 650
- Dose Expansion Phase Group 1: TNBC (Experimental): Participants with locally advanced or metastatic triple negative breast cancer (TNBC), will be administered with the preliminary RP2D identified from the dose exploration part of the study.
  Interventions: Drug: AMG 650
- Dose Expansion Phase Group 2: HGSOC (Experimental): Participants with locally advanced or metastatic high grade serous ovarian cancer (HGSOC), will be administered with the preliminary RP2D identified from the dose exploration part of the study.
  Interventions: Drug: AMG 650

INTERVENTIONS:
Drug: AMG 650 — AMG 650 administered orally as a tablet.

SUMMARY:
To evaluate the safety and tolerability of AMG 650 in adult participants and to determine the maximum tolerated dose (MTD) and/or recommended phase 2 dose (RP2D).

ELIGIBILITY:
Inclusion Criteria:

* Male and female ≥ 18 years old
* Triple Negative Breast Cancer participants only: Participant must have histologically or cytologically confirmed metastatic or locally recurrent estrogen receptor (ER)-negative (<1% by immunohistochemistry [IHC]), progesterone receptor (PR)-negative (<1% IHC) and human epidermal growth factor receptor 2 (Her2)-negative (either fluorescent in situ hybridisation [FISH] negative, 0 or 1+ by IHC, or IHC2+ and FISH negative per ASCO/CAP definition) breast cancer. Participant must be relapsed/refractory to at least one line of systemic chemotherapy in the metastatic setting (excluding neoadjuvant or adjuvant chemotherapies) or intolerant of existing therapy(ies) known to provide clinical benefit or have no other available treatment options. Prior exposure to an immune checkpoint inhibitor is allowed.
* Platinum-Resistant High Grade Serous Ovarian Cancer, primary peritoneal cancer and/or fallopian-tube cancer participants only: Participant must have histologically or cytologically confirmed diagnosis of metastatic or unresectable high grade serous ovarian cancer, with platinum-resistance defined as progression during or within 6 months of a platinum-containing regimen, with no other treatment option available. Prior exposure to platinum-resistant recurrence therapy is allowed.
* Serous Endometrial Cancer participants only (Dose Exploration only): Participant must have histologically or cytologically confirmed diagnosis of metastatic or recurrent serous endometrial cancer, and be relapsed/refractory to at least one line of systemic therapy in the metastatic/recurrent setting or intolerant of existing therapy(ies) known to provide clinical benefit for their condition.
* Participants with advanced or metastatic solid tumor with TP53MUT (Dose Exploration only, as assessed by local testing) that is unresectable and relapsed/refractory to at least one line of systemic chemotherapy or intolerant.
* TNBC participants only (Dose Expansion): Progressed on no more than 3 prior lines of systemic therapy for locally advanced or metastatic disease (not including adjuvant or neo-adjuvant). Systemic therapy with poly ADP ribose polymerase (PARP) inhibitor will be counted as one line of therapy.
* HGSOC participants only (Dose Expansion): Progressed on no more than 5 prior lines of systemic therapy for locally advanced or metastatic disease (not including adjuvant or neo-adjuvant). Systemic therapy with (PARP) inhibitor will be counted as one line of therapy. Induction followed by maintenance will be counted as one line of therapy.

Exclusion Criteria:

* Untreated or symptomatic brain metastases and leptomeningeal disease (exception: benign asymptomatic tumors are permitted).
* Current primary CNS tumor, hematological malignancies or lymphoma.
* Uncontrolled pleural effusions(s), pericardial effusion, or ascites.
* Gastrointestinal (GI) tract disease causing the inability to take oral medication.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2020-03-11 (Actual); Primary Completion 2022-10-24 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Dose Limiting Toxicities (DLTs) | Up to 12 months
Number of Participants with Treatment-emergent Adverse Events (TEAEs) | Up to 24 months
Number of Participants with Serious Adverse Events (SAEs) | Up to 24 months
Number of Participants with Treatment-related Adverse Events | Up to 24 months
Number of Participants Who Experience a Clinically Significant Change from Baseline in Vital Sign Measurement | Up to 24 months
Number of Participants Who Experience a Clinically Significant Change from Baseline in Electrocardiogram (ECGs) Measurement | Up to 24 months
Number of Participants Who Experience a Clinically Significant Change from Baseline in Clinical Laboratory Tests | Up to 24 months

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to 24 months
Duration of Response (DOR) | Up to 24 months
Progression-free Survival (PFS) | Up to 24 months
Clinical Benefit Rate (CBR) | Up to 24 months
Time to Response (TTR) | Up to 24 months
Time to Progression (TTP) | Up to 24 months
Overall Survival (OS) | Up to 24 months
Maximum Plasma Concentration (Cmax) of AMG 650 | Up to 24 months
Time to Maximum Plasma Concentration (Tmax) of AMG 650 | Up to 24 months
Area Under the Plasma Concentration-time Curve (AUC) Over the Dosing Interval for AMG 650 | Up to 24 months

CONTACTS AND LOCATIONS:
Locations (22):
- United States (13):
  - The Angeles Clinic and Research Institute, West Los Angeles Office, Los Angeles, California
  - Sarcoma Oncology Research Center LLC, Santa Monica, California
  - Indiana University, Indianapolis, Indiana
  - Mayo Clinic, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - Roswell Park Cancer Institute, Buffalo, New York
  - Laura and Isaac Perlmutter Cancer Center at New York University Langone, New York, New York
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Texas Oncology - Baylor, Dallas, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
- Australia (2):
  - The Queen Elizabeth Hospital, Woodville South, South Australia
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
- Universitair Ziekenhuis Leuven - Campus Gasthuisberg, Leuven, Belgium
- Canada (2):
  - Cross Cancer Institute, Edmonton, Alberta
  - Princess Margaret Cancer Centre, Toronto, Ontario
- IRCCS Istituto Europeo di Oncologia, Milan, Italy
- Japan (2):
  - Aichi Cancer Center, Nagoya, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa-shi, Chiba
- Hospital General Universitario Gregorio Marañon, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided